CLINICAL TRIAL: NCT04157894
Title: Estimating the Malaria Prevention Impact of New Nets: Observational Analyses to Evaluate the Evidence Generated During Piloted New Net Distributions in Burkina Faso
Status: Completed | Type: Observational
Sponsor: PATH (Other)
Collaborators: Centre national de recherche et de formation sur le paludisme (Other Government); Liverpool School of Tropical Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 1379279-2
Record Dates: First submitted 2019-10-03; First posted 2019-11-08 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-01

CONDITIONS: Malaria
Keywords: Long-lasting insecticidal net; LLIN; Insecticide treated net; ITN; Malaria; Epidemiology; Anthropology; Durability; Cost-effectiveness
MeSH Terms: conditions — Malaria | interventions — milbemycin oxime

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Standard LLIN: This group receives Interceptor ITNs during the mass distribution campaign.
  Interventions: Other: Standard long-lasting insecticidal net
- Chlorfenapyr ITN: This group receives Interceptor G2 ITNs during the mass distribution campaign.
  Interventions: Other: Chlorfenapyr insecticide treated net
- Piperonyl butoxide LLIN: This group receives PBO ITNs during the mass distribution campaign.
  Interventions: Other: Piperonyl butoxide long-lasting insecticidal net

INTERVENTIONS:
Other: Standard long-lasting insecticidal net — Interceptor® (BASF) contains a pyrethroid insecticide
  Other Names: Interceptor®
  Groups: Standard LLIN
Other: Chlorfenapyr insecticide treated net — Interceptor® G2 (BASF) is an ITN containing two active ingredients: Alpha-cypermethrin, a pyrethroid insecticide, and chlorfenapyr, a pyrrole insecticide.
  Other Names: Interceptor G2®
  Groups: Chlorfenapyr ITN
Other: Piperonyl butoxide long-lasting insecticidal net — PermaNet®3.0 (Vestergaard) contains deltamethrin, a pyrethroid insecticide, and piperonyl butoxide, an insecticide synergist.
  Other Names: PermaNet®3.0
  Groups: Piperonyl butoxide LLIN

SUMMARY:
The use of insecticide-treated bed nets (ITN) has contributed to the substantial reduction in malaria cases and deaths. This progress is threatened by increasing resistance commonly used insecticides in mosquito populations. Newly developed, next-generation ITNs using two insecticides or an insecticide synergist and an insecticide are effective against resistant mosquitoes, but large-scale uptake of these nets has been slow due to higher costs and lack of enough evidence to support broad policy recommendations.

This observational study will occur alongside a pilot distribution of next-generation ITNs and collect data over three years on their entomological and epidemiological impact as well as anthropological factors that influence their uptake and use. Data collection will occur in three districts: one receiving dual-active ingredient ITNs, Interceptor® G2 (BASF), one receiving a standard pyrethroid long-lasting insecticidal net (LLIN), Interceptor® (BASF), and one receiving PermaNet®3.0 (Vestergaard) an LLIN containing an insecticide and an insecticide synergist. Data will be collected on malaria vector bionomics, disease epidemiology, and human behaviors in order to help better demonstrate the public health value of next-generation ITNs and to support donors, policymakers, and National Malaria Control Programs in their ITN decision-making and planning processes.

DETAILED DESCRIPTION:
The World Health Organization's (WHO) 2018 World Malaria Report estimates that in 2017, 219 million cases of malaria occurred worldwide resulting in 435,000 deaths, 93% of which occurred in Africa. While this represents a remarkable improvement in comparison with 2000, with malaria deaths having fallen by 40% in Africa, the downward trends in incidence and mortality stalled between 2015 and 2017. This recent failure to maintain the hard-won progress, let alone accelerate progress towards elimination, over the past three years has caused WHO to describe the global fight against malaria as being at a cross roads, calling for increased funding and highlighting the need to develop, optimize, and implement new tools to combat malaria.

Universal coverage of populations at risk with malaria vector control interventions-primarily insecticide treated nets (ITNs) and indoor residual spraying (IRS)-in malaria-endemic countries is a global and national priority because of its fundamental importance for malaria control and elimination. Unfortunately, the effectiveness of these tools is threatened by the emergence and spread of pyrethroid resistance in key mosquito populations, which is now reported in more than 85% of all malaria endemic countries and poses significant risk to the future impact of these tools. Emerging evidence suggests, however, that increasing mosquito mortality-and thereby continuing to reduce malaria transmission-is possible in areas with pyrethroid resistance by introducing new insecticide formulations for IRS and ITNs. For example, Protopopoff et al. showed in Tanzania that the distribution of LLINs with piperonyl butoxide (PBO) plus pyrethroid reduced malaria prevalence by 13% compared to standard pyrethroid-only LLIN distribution (42% vs. 29%; p=0.0011), and Tiono et al., working in Burkina Faso, showed that the distribution of a dual active-ingredient ITN reduced clinical malaria incidence by 22% (Incidence Rate Ratio = 0.88; p=0.04) and potentially infective mosquito bites by 51% (entomological inoculation rate ratio = 0.49; p<0.0001) compared to the distribution of a standard pyrethroid-only LLIN.

While there is evidence that standard LLINs can continue to provide effective personal protection to regular net users in regions with resistant vector populations, new classes of ITNs developed to perform against pyrethroid-resistant mosquitoes have been developed, with early trials and modelling suggesting that they may provide superior protective efficacy against malaria in areas with pyrethroid-resistant vectors. Access to these new resistance-breaking ITNs is restricted by need for efficacy data for continuing policy recommendations, high prices, lack of evidence of cost effectiveness compared to pyrethroid-only LLINs, and consequent poor demand in an uncertain market. Interceptor® G2 (IG2) (BASF), a new type of ITN consisting of two active ingredients including a mixture of a pyrethroid (alpha-cypermethrin) and a pyrrole (chlorfenapyr) insecticide, recently achieved WHO prequalification listing demonstrating that it performs to the thresholds required of pyrethroid-only LLINs and has no known specific side effects. While the IG2 ITN has been subsequently registered and approved for use in Burkina Faso based on this WHO listing the Roll Back Malaria Vector Control Advisory Group guidance indicates that dual active ingredient ITNs will require further epidemiological evidence before policy recommendations are made for their use in preference to pyrethroid-only LLINs in certain settings.

The Global Fund and Unitaid have developed a market shaping program for IG2 and other ITNs with novel insecticide formulations. Evidence on the efficacy of IG2s will be generated by the project through two randomized control trials taking place in Benin and Tanzania. In addition, through this program, these next-generation ITNs will be made available to countries for incorporation into their national distribution programs as pilot distributions with the aim of determining real-world effectiveness and cost-effectiveness in different contexts. In addition to the pilot distribution of IG2s taking place in Burkina Faso, three other countries will be piloting IG2s as part of the New Nets project: Mali, Mozambique, and Rwanda. This research will utilize these pilot distributions to understand the cost-effectiveness of the new ITNs in the chosen settings. The NMCP in Burkina Faso, in discussion with the Global Fund, chose to incorporate IG2 ITNs into the upcoming 2019 mass distribution campaign. This study covers gathering information to determine the public health impact of the IG2 ITNs in Burkina Faso, in comparison to sites that will receive standard pyrethroid-only LLINs or PBO LLINs during the mass campaign. The aim of this research is to better understand the effectiveness and cost effectiveness of IG2 ITNs in Burkina Faso and to collect data on community uptake of the ITNs. During the upcoming pilot implementation, entomological, epidemiological, and anthropological data will be collected in up to three study districts, one that will receive IG2 ITNs, one comparator district that will receive standard LLINs, and one additional comparator district that will receive PBO LLINs. Data will be analyzed, and results disseminated to support the NMCP, donors, policymakers, and other national and regional stakeholders in their ITN decision-making and planning processes.

As part of the New Nets Project initiative to catalyze the market introduction of next-generation ITNs, Burkina Faso will be piloting the deployment of next-generation ITNs in selected districts where enhanced surveillance activities will be used to support observational impact analyses. This study aims to provide National Malaria Control Programs (NMCP), international donors and other key stake holders with evidence on the impact next-generation ITNs on malaria burden. The decision on which type of ITNs to be distributed and where to distribute them were all made by the national control program with the support of international donors. These ITNs have gone through the country's appropriate registration process prior to their purchase and delivery in-country. This observational study is opportunistic in the sense that it is taking advantage of the decision of the national program to distribute the different ITNs (standard and next-generation) in different districts to evaluate their impact on malaria burden.

In these districts, epidemiological, entomological, and anthropological data will be collected with the primary goal of evaluating the effectiveness and cost-effectiveness of deploying next-generation ITNs. Each component specifically aims to:

* Epidemiological component - measure the epidemiological impact of the new IG2 ITNs, standard LLINs, and PBO LLINs in real deployment scenarios through observational studies. These studies will compare trends in (1) malaria case incidence rates passively reported to the national health system (passive case detection, PCD) and (2) malaria infection prevalence, measured through Rapid Diagnostic Tests (RDTs), in children 6 to 59 months of age from annual cross-sectional surveys during peak transmission periods.
* Entomological component - evaluate the impact of IG2 ITNs on vector populations and biting rates, compared to standard and PBO LLINs, through national mosquito surveillance data that will measure trends in species- specific (1) adult vector densities (2) indoor and outdoor human landing rates (3) estimated entomological inoculation rates and (4) insecticide resistance patterns.
* Anthropological component - map the social determinants of impact for IG2 LLINs and determine transmission risk defined as the intersection between time at risk of mosquito blood feeding and human activities not under protection of an ITN, through gathering evidence on LLIN uptake and usage. The collection of reliable data on such patterns, both indoors and outdoors, becomes thus an essential component of the evaluation of the ITN pilots for both modeling and contextual analysis of impact.
* Costing and cost-effectiveness component - estimate the cost and cost-effectiveness of IG2 ITNs in southwest Burkina Faso through data on the price of the product, delivery and deployment costs, and product effectiveness based on case incidence rates measured during the epidemiological component of this study. Additionally, mean costs per case averted that might occur in other contexts will be modeled and incorporated into the cost-effectiveness evaluations.

ELIGIBILITY:
Inclusion Criteria:

* Passive data collection: All suspected malaria cases (fevers) that self-present to the national health system and are counted in the district health surveillance systems.
* Cross-sectional survey: Households in the district with a family member from the target age group.

  * Residents of the household visited.
  * Questionnaire: parent or guardian giving written informed consent (cross-sectional).
  * Malaria screening: child aged 6 to 59 months from the above consenting household.
* Individuals of box sexes, not belonging to vulnerable categories (those with cognitive impairment or other person for whom full and open consent cannot be guaranteed) (Key informant interviews, focus group discussions, and participant observations).
* Individuals 20 years old and above (key informant interviews, focus group discussions, participant observations).
* Individuals of both sexes regardless of age (structured observations).

Exclusion Criteria:

* District non-residents.
* Malaria screening: history of recent (within one month) malaria infection or treatment with anti-malarial medication (cross-sectional).
* Parents or guardians who have not yet reached age of consent (20 years) and their children will not be included in study activities requiring consent.
* Individuals belonging to vulnerable categories (key informant interviews, focus group discussions, participant observations).
* Individuals unwilling and/or unable of giving consent (key informant interviews, focus group discussions, participant observations).
* Individuals below age of consent (20 years) (key informant interviews, focus group discussions, participant observations)
* Heads of households unwilling and/or unable of giving consent (structured observations)
* Individuals who do not wish to be included in observations will be excluded (structured observations)

Min Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Cohorts will be selected from the population of five districts, Banfora, Gaoua, Orodara, Nouna, and Tougan, that will receive nets as part of the Burkina Faso mass distribution campaign of ITNs. The districts have similar malaria transmission dynamics. Routine data provided by in-country stakeholders show that these districts are comparable in underlying malaria prevalence, incidence, vector species composition, and insecticide resistance status, as well as general climate and geographic similarities. The three southern districts (Orodara, Gaoua, Banfora) will receive enhanced data collection support, and the two northern districts (Nouna and Tougan) will be analyzed using routine health system data. Limit: 1000 characters.
Sampling Method: Probability Sample
Enrollment: 5606 (Actual)
Dates: Start 2019-07-07 (Actual); Primary Completion 2022-07-06 (Actual); Study Completion 2022-07-06 (Actual)

PRIMARY OUTCOMES:
Cumulative malaria incidence | July 2019 to December 2022, monthly
  Malaria incidence measured through passive case detection at health facilities in each district. This measure accounts for symptomatic cases self-reporting to the formal health system for care.

SECONDARY OUTCOMES:
Vector species composition | July 2019 to December 2022, monthly
  All Anopheles mosquitoes sampled during Centers for Disease Control and Prevention light traps (CDCLT) and human landing collections (HLC) will be identified morphologically to species group
Species-specific population densities | July 2019 to December 2022, monthly
  Based on Anopheles mosquitoes sampled during CDCLT
Biting behaviors | July 2019 to December 2022, monthly
  Based on Anopheles mosquitoes sampled during CDCLT
Estimated entomological inoculation rates | July 2019 to December 2022, monthly
  Based on Anopheles mosquitoes sampled during CDCLT and HLC
Insecticide resistance profile | July 2019 to December 2022, monthly
  Measurement of kdr and ace-1 mutation frequencies, WHO tube bioassays at minimum and CDC bottle bioassays to characterize insecticide resistance intensity
Parasite prevalence in children 6-59 months | July 2019, July 2020, July 2021, July 2022
  Prevalence calculated from cross-sectional surveys conducted during the peak transmission season.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Wagman, PhD, Principal Investigator — PATH; Sagnon NFalé, MD, Principal Investigator — Centre national de recherche et de formation sur le paludisme
Locations (1):
- Centre National de Recherche et de Formation sur le Paludisme, Ouagadougou, Burkina Faso

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alonso P, Noor AM. The global fight against malaria is at crossroads. Lancet. 2017 Dec 9;390(10112):2532-2534. doi: 10.1016/S0140-6736(17)33080-5. Epub 2017 Nov 29. No abstract available. PMID 29195688
- [Background] Badolo A, Traore A, Jones CM, Sanou A, Flood L, Guelbeogo WM, Ranson H, Sagnon N. Three years of insecticide resistance monitoring in Anopheles gambiae in Burkina Faso: resistance on the rise? Malar J. 2012 Jul 16;11:232. doi: 10.1186/1475-2875-11-232. PMID 22799568
- [Background] Bass C, Nikou D, Donnelly MJ, Williamson MS, Ranson H, Ball A, Vontas J, Field LM. Detection of knockdown resistance (kdr) mutations in Anopheles gambiae: a comparison of two new high-throughput assays with existing methods. Malar J. 2007 Aug 13;6:111. doi: 10.1186/1475-2875-6-111. PMID 17697325
- [Background] Bayili K, N'do S, Namountougou M, Sanou R, Ouattara A, Dabire RK, Ouedraogo AG, Malone D, Diabate A. Evaluation of efficacy of Interceptor(R) G2, a long-lasting insecticide net coated with a mixture of chlorfenapyr and alpha-cypermethrin, against pyrethroid resistant Anopheles gambiae s.l. in Burkina Faso. Malar J. 2017 May 8;16(1):190. doi: 10.1186/s12936-017-1846-4. PMID 28482891
- [Background] Bhatt S, Weiss DJ, Cameron E, Bisanzio D, Mappin B, Dalrymple U, Battle K, Moyes CL, Henry A, Eckhoff PA, Wenger EA, Briet O, Penny MA, Smith TA, Bennett A, Yukich J, Eisele TP, Griffin JT, Fergus CA, Lynch M, Lindgren F, Cohen JM, Murray CLJ, Smith DL, Hay SI, Cibulskis RE, Gething PW. The effect of malaria control on Plasmodium falciparum in Africa between 2000 and 2015. Nature. 2015 Oct 8;526(7572):207-211. doi: 10.1038/nature15535. Epub 2015 Sep 16. PMID 26375008
- See also: Ben-Shlomo Y, Brookes S, Hickman M. Lecture Notes: Epidemiology, Evidence-based Medicine and Public Health. — https://www.wiley.com/en-us/Lecture+Notes%3A+Epidemiology%2C+Evidence+based+Medicine+and+Public+Health%2C+6th+Edition-p-9781444334784
- See also: Bernard, HR. Research Methods in Anthropology: Qualitative and Quantitative Approaches. 4th — http://www.dphu.org/uploads/attachements/books/books_476_0.pdf